CLINICAL TRIAL: NCT02660320
Title: Comparison of the Efficacy of Micro-holes vs. Laser-assisted Dermabrasion, for Repigmenting in Vitiligo Skin
Acronym: Dermabrasion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-PP-09
Record Dates: First submitted 2016-01-04; First posted 2016-01-21 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2018-01

CONDITIONS: Vitiligo - Macular Depigmentation
MeSH Terms: interventions — Dermabrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermabrasion (Active Comparator): Dermabrasion using dermaroller: The dermaroller is applied on the treated areas, this dermabrasion technique is based on micro holes performed using 540 micro needles (200µm depth) which should allow the penetration of the suspension cells or hyaluronic acid alone. Twelve passages will be performed on the treated area in order to achieve 60% of coverage.
  Interventions: Device: Dermabrasion
- Laser (Placebo Comparator): To prepare the graft recipient site, the upper layer of epidermis is removed by superficial dermabrasion using Erbium or CO2 ablative laser. The test area is ready to receive suspension cells when the dermis will appeared. The cells suspension will be applied on the wound.
  Interventions: Device: Laser placebo

INTERVENTIONS:
Device: Dermabrasion — Preparing the graft bed before epidermal cell suspension The epidermis can be removed using ablative CO2 or Erbium laser. We will assess the efficacy of using instead micro-needles to create micro-holes that will allow the melanocytes to reach the lower layers of the epidermis and thus repigment the lesional skin.
  Arms: Dermabrasion
Device: Laser placebo — The epidermis can be removed using ablative CO2 or Erbium laser. We will assess the efficacy of using instead micro-needles to create micro-holes that will allow the melanocytes to reach the lower layers of the epidermis and thus repigment the lesional skin.
  Arms: Laser

SUMMARY:
Principal objective: To compare the efficacy of laser-assisted dermabrasion + autologous epidermal cells suspension grafting versus dermabrasion using micro-needling technique + autologous epidermal cells suspension grafting and dermabrasion using micro-needling technique + placebo suspension grafting in stable vitiligo.

A total of 10 patients with stable non-segmental vitiligo will be included in the ITT population.

In each patient, three separate test areas will be selected in the same part of the body.

One area will be pre-treated with dermaroller and receive the hyaluronic acid suspension alone and the two others will receive the epidermal cell suspension in hyaluronic acid after pre-treatment either with dermaroller or laser-assisted dermabrasion, each patient being his own control.

Targeted phototherapy with excimer lamp (308 nMm) will be applied on all test areas 1 week after cell grafting.

DETAILED DESCRIPTION:
Condition Stable lesion of Vitiligo of adulthood

Background Laser-assisted dermabrasion is the gold standard for preparing the grafting bed of epidermal suspension but it requires a technical platform and a trained physician. Side effects are not uncommon. We have demonstrated in an ex vivo study that micro-needles create holes in the epidermis allowing cells to reach the lower layers of the epidermis. We hypothesize that the use of micro-needles could be an effective and easy technique for preparing the grafting bed for epidermal suspensions.

Objectives Principal objective: To compare the efficacy of laser-assisted dermabrasion + autologous epidermal cells suspension grafting versus dermabrasion using micro-needling technique + autologous epidermal cells suspension grafting and dermabrasion using micro-needling technique + placebo suspension grafting in stable vitiligo.

The secondary objectives are

1. To evaluate and compare the tolerability of the distinct procedures
2. To evaluate the global satisfaction of patient and the willingness to reproduce the procedure for treating other areas
3. To evaluate the contrast between treated skin and perilesional area

Methods Prospective, multicentre, randomized, controlled, blind assessor trial.

Inclusion criteria

* Men and women aged over 18 years old with a diagnosis of non-segmental lesions that has been stable over three months
* The minimum distance between the normal pigmented skin and the test area should preferably be at least 0.5 cm.
* For each patient the lesions are located on the same area (either chest, back, legs or arms)
* The lesion area must be: 2cm2 < lesion<50cm2
* Treatment resistant areas (failure of at least one medical procedure topical tacrolimus or topical steroids for 6 months).
* Absence of infected lesion
* Lesions stable for at least one year

Exclusion criteria Hypersensibility to local anaesthetics or one of the components of the device (trypsin, hyaluronic acid)

* Indication against biopsies
* Patient with a history of melanoma
* Positive serology (ongoing serious systemic disease, herpes, HIV, hepatitis B and C)
* History of keloidal scars and presence of Koebner's phenomenon (type 1 and type 2b)
* Infected lesion
* Patient with concomitant photosensitizing treatment
* Age <18 years
* Major deprived of their freedom by administrative or legal decision, or being the subject of a legal protection measure, or out of state to express their consent
* Pregnant,delivering or lactating patients. For the women childbearing potential, a urinary pregnancy test will be done and effective contraception will be expected.

Interventions After inclusion visit, randomization will occur during visit 1, the day of the surgery to determine which lesion will be treated by dermaroller+hyaluronic acid, dermaroller+VITICELL® or laser-assisted dermabrasion+VITICELL®.

Dermabrasion procedures:

Three test areas will be selected on the same part of body. Each lesion will respectively treated by:

* Dermaroller + hyaluronic acid + phototherapy
* Dermaroller + VITICELL® + phototherapy
* Laser + VITICELL® + phototherapy

Dermabrasion using laser:

To prepare the graft recipient site, the upper layer of epidermis is removed by superficial dermabrasion using Erbium or CO2 ablative laser. The test area is ready to receive suspension cells when the dermis will appeared. The cells suspension will be applied on the wound.

Dermabrasion using dermaroller: The dermaroller is applied on the treated areas, this dermabrasion technique is based on micro holes performed using 540 micro needles (200µm depth) which should allow the penetration of the suspension cells or hyaluronic acid alone. Twelve passages will be performed on the treated area in order to achieve 60% of coverage.

VITICELL® treated area:

A small sample of skin (biopsy) will be collected from the gluteal area. The biopsy will be measured 4 cm2 (2x2cm) systematically. While the investigator is preparing the areas to be treated, the skin will be placed into the VITICELL® kit by other heath professional. The VITICELL® kit will transform the patient's collected skin into a cellular suspension. The suspension of epidermal cells is then applied (100µL per cm2) onto the 2 selected lesions/areas after dermabrasion with dermaroller or laser.

Hyaluronic acid with PBS treated area:

The suspension of hyaluronic acid is applied (100 µL/cm2) onto the selected lesion after dermabrasion with dermaroller.

Following the surgery, the treated area and biopsy site will be covered with a dressing and must be protected from direct sun and physical impact for a period of 6 -7days. After this period the dressing will be removed.

Phototherapy:

The phototherapy will begin a week after cells grafting and will be used 2 times a week for all the treatment duration.

The ultraviolet (UV) spectrum has been used on test areas. These different wavelength will promote melanogenesis and melanocyte proliferation on graft side.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years old with a diagnosis of non-segmental lesions that has been stable over three months
* The minimum distance between the normal pigmented skin and the test area should preferably be at least 0.5 cm.
* For each patient the lesions are located on the same area (either chest, back, legs or arms)
* The lesion area must be: 2cm2 < lesion<50cm2
* Treatment resistant areas (failure of at least one medical procedure topical tacrolimus or topical steroids for 6 months).
* Absence of infected lesion
* Lesions stable for at least one year

Exclusion Criteria:

* Hypersensibility to local anaesthetics or one of the components of the device (trypsin, hyaluronic acid)
* Indication against biopsies
* Patient with a history of melanoma
* Positive serology (ongoing serious systemic disease, herpes, HIV, hepatitis B and C)
* History of keloidal scars and presence of Koebner's phenomenon (type 1 and type 2b)
* Infected lesion
* Patient with concomitant photosensitizing treatment
* Age <18 years
* Major deprived of their freedom by administrative or legal decision, or being the subject of a legal protection measure, or out of state to express their consent
* Pregnant,delivering or lactating patients. For the women childbearing potential, a urinary pregnancy test will be done and effective contraception will be expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Rate of repigmentation lesions | at 3 months
  Rate of repigmentation lesions at 3 months

SECONDARY OUTCOMES:
Global satisfaction expressed by the patient | at 3 months
  Global satisfaction expressed by the patient per treated area at the end of the treatment
EVA scale | During the procedure
  Pain expressed by the patient during the procedure (EVA scale)
-Contrast between treated and perilesional area (Nottingham scale) | at 3 months
  Contrast between treated and perilesional area (Nottingham scale)

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Dermatology, CHU de Nice
Locations (3):
- France (3):
  - CHU de Nice, Nice, Alpes-Maritimes
  - CHU de Bordeaux, Bordeaux
  - CH Creteil, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided